CLINICAL TRIAL: NCT04315051
Title: Clinical Trial Protocol DBI-204 Double-Blind, Randomized, Placebo Controlled Trial of the Safety and Efficacy of DBI-001 Gel in Patients With Interdigital Tinea Pedis
Brief Title: A Trial of Safety/Efficacy of Test Article in Patients With Interdigital T. Pedis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid- 19 has shut the clinic
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DBI-204
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-02

CONDITIONS: Interdigital Tinea Pedis

STUDY DESIGN:
Intervention Model Description: A Double-Blind, Randomized, Placebo Controlled trial of the Safety and Efficacy of DBI-001 Gel in patients with interdigital T. pedis. Test articles will be applied by subjects once daily at bedtime for a period of four (4) weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Gel (Placebo Comparator): Placebo gel daily application for 4 weeks
  Interventions: Other: Placebo Gel
- Cohort 1 (Active Comparator): DBI-001 Gel daily application for 4 weeks
  Interventions: Drug: Cohort 1 J. Lividum

INTERVENTIONS:
Drug: Cohort 1 J. Lividum — Subject to apply DBI-001 Gel on each foot covering all web spaces, the plantar and lateral aspects, toes and toenails
  Arms: Cohort 1
Other: Placebo Gel — Subject to apply Placebo Gel daily on each foot covering all web spaces, the plantar and lateral aspects, toes and toenails.
  Arms: Placebo Gel

SUMMARY:
Placebo Controlled Trial of the Safety and Efficacy of DBI-001 in Patients with Interdigital Tinea pedis (T. pedis)

DETAILED DESCRIPTION:
Double-Blind, Randomized, Placebo Controlled Trial of the Safety and Efficacy of DBI-001 Gel in Patients with Interdigital Tinea pedis (T. pedis). The primary objective is to observe the antimicrobial effect of a daily application of DBI-001Gel for 4 weeks in patients with interdigital T. pedis based on the change from culture positive for a dermatophyte to culture negative as determined by routine mycology culture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be included in the study:

  1. A signed approved informed consent form by Institutional Review Board/Independent Ethics Committee.
  2. A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of subject's individually identifiable health information.
  3. Male or Female Subjects of any race 18 years of age and older.
  4. Women patients of child-bearing potential must: a. Have negative urine pregnancy tests prior to study treatment to rule out pregnancy, and b. Use at least one method of birth control that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner for the duration of study participation.
  5. Subjects with a clinical diagnosis of interdigital T. pedis T. pedis interdigital defined as lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin).
  6. Provisionally confirmed diagnosis at screening by a positive potassium hydroxide (KOH) wet mount at the clinical site.
  7. A positive dermatophyte culture from the sample obtained at the screening visit.
  8. The sum of the clinical signs and symptoms scores of at least one web space (Target web space) is at least 4 using the Grading of Signs and Symptoms of T. pedis including a minimum score of at least 2 for erythema AND a minimum score of 2 for either scaling/fissures or pruritus/burning (on a scale of 0-3, where 2 indicates moderate severity).
  9. Target web space should have adequate amount of leading-edge scale to provide enough scale for KOH, fungal culture and molecular diagnostics.

     Exclusion Criteria:

     Subjects with the following will be excluded from this study:

  <!-- -->

  1. Females who are pregnant, planning a pregnancy, breastfeeding or have a positive pregnancy test at the site.
  2. Any dermatological conditions that could interfere with clinical evaluations.
  3. The clinical diagnosis of moccasin T. pedis.
  4. Any underlying disease(s) or some other dermatological condition that requires the use of interfering topical or systemic therapy.
  5. Subjects that have not undergone the specified washout period(s) or subjects who require the concurrent use of specific topical medications applied to the foot.
  6. Subjects that have not undergone the washout periods for systemic medications or who require the use of specific systemic medications.
  7. Treatment of any type of cancer within the last 6 months.
  8. History of any significant internal disease (which contraindicates use of live microbiome e.g. leukemia, liver failure, cardiovascular disease).
  9. Subjects who are known to be allergic to any of the Test Article(s) or any components in the Test Article(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
  10. AIDS or AIDS related complex by medical history.
  11. Known or suspected immune suppressive medications or diseases.
  12. Diabetes mellitus Type I or II by medical history.
  13. Peripheral vascular disease based on medical history.
  14. Any subject not able to meet the study attendance requirements.
  15. Subjects who have participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
From Culture Positive to Culture Negative | Baseline (Day 1) to Day 28
  Antimicrobial effect. Effect will be measured by change from culture positive for dermatophyte to culture negative as determined by routine mycology culture.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Blanco, MD, Study Director — Instituto Dermatologico y Cirugia de Piel
Locations (1):
- Instituto Dermatologico y Cirugia de Piel, Santo Domingo, Dominican Republic